CLINICAL TRIAL: NCT07252453
Title: Comparison of Carbamazepine and Oxcarbazepine In the Treatment of Trigeminal Neuralgia
Brief Title: Comparison b/w Carbamazepine vs Oxcarbazepine in Treatment of Trigeminal Neuralgia
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbasi Shaheed Hospital (Other)
Responsible Party: Principal Investigator, Sikandar Zaidi, Resident (PG R3), Abbasi Shaheed Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB/KMDC/KMU/128/2025
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Trigeminal Neuralgia
Keywords: TGN; carbamazepine; oxcarbazepine
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Carbamazepine; Oxcarbazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Carbamazepine group (Active Comparator): In this group participants has been prescribed with carbamazepine which is conventional drug for trigeminal neuralgia management
  Interventions: Drug: Carbamazepine
- Oxcarbazepine group (Active Comparator): In this group participants has been prescribed with oxcarbazepine which is new FDA approved drug for TGN management
  Interventions: Drug: oxcarbazepine

INTERVENTIONS:
Drug: Carbamazepine — Carbamazepine is a conventional drug used to treat trigeminal neuralgia. It primarily works by blocking voltage-gated sodium channels in nerve cells, which prevents rapid and repetitive firing of action potentials and reduces abnormal electrical activity in the brain.
  Arms: Carbamazepine group
Drug: oxcarbazepine — Oxcarbazepine is comparatively new approved drug in the treatment of TGN. Oxcarbazepine is a prodrug that is rapidly converted to its active metabolite, (monohydroxy metabolite or MHD). This active form works by blocking voltage-sensitive sodium channels in the brain, which stabilizes over-excited nerve membranes and prevents the rapid spread of abnormal electrical activity
  Arms: Oxcarbazepine group

SUMMARY:
In this Study investigator is comparing the effectiveness and outcomes of two drugs used un the treatment of trigeminal neuralgia , Carbamazepine vs Oxcarbazepine

DETAILED DESCRIPTION:
In this open pilot open label randomized controlled trial, Investigator is comparing the effectiveness and outcomes of two drugs used un the treatment of trigeminal neuralgia, Carbamazepine vs Oxcarbazepine , hypothesis would be that oxcarbazepine has equal or better outcomes comparatively with less side effects

ELIGIBILITY:
* Inclusion Criteria:

  * Age 18-60 years
  * Either gender
  * TGN diagnosis for ≥2 weeks (according to ICHD-3 criteria¹)

Exclusion Criteria [Expanded]:

* Other cranial neuralgias
* Prior surgical treatment for TN
* Hepatic/renal dysfunction
* Epilepsy
* Pregnant/lactating women
* Drug allergy or intolerance
* [Expanded] Uncontrolled hypertension
* [Expanded] Psychiatric disorders

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain relief for TGN | Two months
  Pain relief for Trigeminal neuralgia will be assessed define as complete resolution of symptoms (PAIN) , after prescribing both drugs to each individual group, Pain relief will be assessed using visual analogue scale (VAS SCORE) , which is designated by number 1 to 10, in which 1 means NO PAIN, and 10 means SEVERE PAIN. Annexure will be provided to each participant which includes study consent, demographic details, medical history in relevance with inclusion and exclusion criteria, side effects , LFTs values and printed Visual Analogue Scale on the very same document.

SECONDARY OUTCOMES:
Side effects | Two months
  Side effects of each drug will be compared including hepatotoxicity through liver functional tests, and other effects including nausea tolerability, dizziness etc. Annexure will be provided to each group participants ( same as mentioned in primary outcome section) ,which includes side effects column specifically Liver Functional Test results including both baselines values ( during the start of treatment ) and final results( at the end of treatment) and comparison will be made between the two drugs regarding side effects specifically hepatotoxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.SUFYAN AHMED, FCPS, Study Chair — KARACHI METROPOLITAN UNIVERSITY/ ABBASI SHAHEED HOSPITAL
Locations (1):
- Abbassi Shaheed hospital Facio-Maxillary Department, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcomes
Supporting Information: Study Protocol
Time Frame: As soon as the article will get published , probably from next year (2027)
Access Criteria: PUBLIC

REFERENCES:
- [Background] 1. International Headache Society. The International Classification of Headache Disorders (ICHD-3) - online edition, updated 2023. Available at: https://ichd-3.org
- See also: Related Info — https://ichd-3.org